CLINICAL TRIAL: NCT05709795
Title: CTI Ablation Guided by Omnipolar Wave Speed and Voltage Maps to Diminish RF and Fluoroscopy Times
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Ermengol Vallès, Doctor, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMNIFLUTTER
Record Dates: First submitted 2022-11-04; First posted 2023-02-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Flutter

STUDY DESIGN:
Intervention Model Description: Prospective randomized multicentric
Who Masked: Participant
Masking Description: Patient won´t know what strategy has been followed to achieve CTI block
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Confluent areas (Experimental): Ablation first of confluent areas of low wave speed and high voltage in the CTI
  Interventions: Procedure: Confluent areas
- Wave Speed (Experimental): Ablation first of areas of low wave speed in the CTI
  Interventions: Procedure: Wave Speed
- Voltage (Active Comparator): Ablation first of areas of high voltage in the CTI
  Interventions: Procedure: Voltage
- CTI line (Active Comparator): Direct CTI line performance (gold standard)
  Interventions: Procedure: CTI line

INTERVENTIONS:
Procedure: Confluent areas — Use of omnipolar technology to guide CTI ablation in sites with both low wave speed and high voltage. If not successful then ablation of low wave speed sites. If not successful then ablation of high voltage sites. If not successful then CTI line (gold standard)
  Other Names: Omnipolar; HD Grid catheter
  Arms: Confluent areas
Procedure: Wave Speed — Use of omnipolar technology to guide CTI ablation in sites with low wave speed. If not successful then ablation of sites with both low wave speed and high voltage. If not successful then ablation of high voltage sites. If not successful then CTI line (gold standard)
  Arms: Wave Speed
Procedure: Voltage — Use of omnipolar technology to guide CTI ablation in sites with high voltage. If not successful then ablation of sites with both low wave speed and high voltage. If not successful then ablation of low wave speed sites. If not successful then CTI line (gold standard)
  Arms: Voltage
Procedure: CTI line — Do not use omnipolar information. CTI line performance
  Arms: CTI line

SUMMARY:
Prospective randomized study involving patients with typical flutter (TF) undergoing cavo-tricuspid isthmus (CTI) radiofrequency ablation. The aim is to compare the results of 3 different new ablation strategies using Omnipolar technology to classic linear ablation.

The investigators´ aim is to compare the effectiveness, safety and procedure times of CTI ablation with 3 different strategies using the Ensite X navigator in magnetic mode with Omnipolar technology and HDGrid catheter to optimize radiofrequency (RF) and fluoroscopy times with classical linear ablation.

The number of patients needed to prove the investigators´ hypothesis is of at least 50 per group (total of 200 prospective patients

DETAILED DESCRIPTION:
Background Ablation procedures for CTI-dependent TF have classically been guided by fluoroscopy and intracavitary electrograms from diagnostic catheters placed in the right atrium (RA), the coronary sinus (CS) and the CTI (ablation catheter). Over the last few years, the use of navigators has increased considerably not only for complex procedures, but also for simple procedures, with the aim of reducing and even completely eliminating irradiation to both the patient and the operator (1). The investigators´ group is looking to characterize the high voltage and the low velocity regions in the CTI to minimize the procedure times. This has been addressed in a recent observational study with very good results.

Rationale There is increasing evidence of the benefits using 3D-systems not only to diminish fluoroscopy, but also to guide ablation targeting high voltage areas in the CTI (2-5). It is well known also the existence of low speed areas in the CTI, facilitating the presence of reentrant circuits (6,7). Currently, the investigators´ center performs all CTI ablation procedures using a 3D-navigator system, mostly with zero or minimal fluoroscopy. The investigators´ group has carried out a preliminary study with 13 patients to assess the effectiveness of CTI ablation with the use of the Ensite X navigator in magnetic mode with Omnipolar technology and HDGrid catheter. In this observational study the investigators were able to characterize the high voltage and the low velocity regions in the CTI to minimize the RF lesions and procedure times. Acute bidirectional block was achieved in 100% of patients with an average fluoroscopy time of 1 ± 2 min (77% patients with zero fluoroscopy) and an average RF time of 5,7 ± 3,2 min (38% below 3 min). This results were significantly lower than results obtained with classical linear ablation: median fluoroscopy time 19.3 min, IQR 12.9 to 36.4 min, median fluoroscopy dose 3520.7 cGycm(2), IQR 1700.0 to 6709.0 cGycm(2).

From the investigators´ point of view this observational study, together with previous evidence justify a randomized study in order to confirm our hypothesis:

Hypothesis Omnipolar technology is able to guide the ablation procedure minimizing both the RF time and the fluoroscopy time (compared to linear ablation) by targeting only the critical regions on the CTI. Therefore Omnipolar technology will diminish RF time and fluoroscopy time/exposition compared to classical CTI ablation, and by means of this the investigators expect an inferior complications rate. Importantly acute success rate and 6 months follow-up recurrences rate will remain similar.

OBJECTIVES

* Primary objectives: to optimize procedure times of CTI ablation with 3 different strategies based in voltage and/or conduction velocity maps using the Ensite X navigator in magnetic mode with Omnipolar technology and HDGrid catheter compared to classical linear ablation.

  o Specific objectives: Fluoroscopy time, radiofrequency time, radiation dose, percentage of zero-fluoroscopy procedures, acute efficacy, complications rate.
* Secondary objectives: to increase the effectiveness of CTI ablation with 3 different strategies based in voltage and/or conduction velocity maps using the Ensite X navigator in magnetic mode with Omnipolar technology and HDGrid catheter compared to classical linear ablation.

  * Specific objectives: Recurrences rate at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to CTI ablation for TF
* Age above 18 years

Exclusion Criteria:

• Life expectancy of <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Radiofrequency time | 24 hours
  Amount of Radiofrequency needed to achieve complete CTI block (acute success)
Fluoroscopy time | 24 hours
  Amount of Fluroscopy time needed to achieve complete CTI block (acute success)
Radiation dose | 24 hours
  Amount of Radiation dose needed to achieve complete CTI block (acute success)
Zero Fluoroscopy | 24 hours
  Percentage of patients performed without the use of fluoroscopy
Acute efficay | 24 hours
  Percentage of acute succeess (complete block of the CTI)
Complications | 2 months
  Percentage of procedural complications

SECONDARY OUTCOMES:
Flutter recurrences | 6 months
  Percentage of recurrences of typical flutter at 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ermengol Valles, Principal Investigator — Hospital del Mar
Locations (2):
- Spain (2):
  - Hospital Germans Tries, Badalona, Barcelona
  - Hospital del Mar, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
RedCap database and randomization tool
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available by the study initiation, on March 2023, and until the publication